CLINICAL TRIAL: NCT01942694
Title: Vitamin D and Type 2 Diabetes Study
Acronym: D2d
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Office of Dietary Supplements (ODS) (NIH); American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U01DK098245 (NIH); U01DK098245 (NIH); NCT02015052 (obsolete NCT alias); NCT02239471 (obsolete NCT alias)
Record Dates: First submitted 2013-08-09; First posted 2013-09-16 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Prediabetes; Type 2 Diabetes
Keywords: Prediabetes; Vitamin D
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2 | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): One pill daily
  Interventions: Other: Placebo
- Vitamin D (Cholecalciferol) (Active Comparator): One vitamin D pill daily
  Interventions: Dietary Supplement: Vitamin D (Cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D (Cholecalciferol) — Vitamin D (Cholecalciferol) 4000 IU, administered as 1 soft-gel pill daily by mouth.
  Arms: Vitamin D (Cholecalciferol)
Other: Placebo — Administered as one soft-gel pill daily by mouth
  Arms: Placebo

SUMMARY:
The goal of the Vitamin D and type 2 diabetes (D2d) study is to determine if vitamin D supplementation works to delay the onset of type 2 diabetes in people at risk for the disease and to gain a better understand how vitamin D affects glucose (sugar) metabolism.

DETAILED DESCRIPTION:
The goal of the Vitamin D and type 2 diabetes (D2d) study is to determine if vitamin D supplementation works to delay the onset of type 2 diabetes in people at risk for the disease and to gain a better understand how vitamin D affects glucose (sugar) metabolism. Researchers at US sites will enroll people with pre-diabetes (people who have higher than normal blood glucose level but not high enough to meet the diagnosis of diabetes). The study will enroll participants over approximately 2 years and participants will be followed for approximately 3 years. Participants will receive either Vitamin D or a placebo by chance. Participants will take 1 pill a day for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-diabetes ("at increased risk for diabetes") defined by meeting 2-out-of-3 of the following glycemic criteria at the baseline visit:

   1. Fasting plasma glucose (FPG) 100-125 mg/dL
   2. 2-hour plasma glucose (2hPG) 140-199 mg/dL
   3. Hemoglobin A1c (HbA1c) 5.7-6.4%
2. Age ≥ 30 years .(≥25 years for people of the following races: American-Indian, Alaska Native, Native Hawaiian or Other Pacific Islander).
3. Body Mass Index ≥ 24.0 (22.5 for Asians) and ≤ 42.0 kg/m2
4. Provision of signed and dated written informed consent prior to any study procedures.

Major Exclusion Criteria:

1. Diabetes based on either of the following criteria:

   1. History (past 1 year) of hypoglycemic pharmacotherapy (oral or injectable medication approved by the FDA for type 2 diabetes), used for any condition (e.g. pre-diabetes, diabetes, polycystic ovarian syndrome.
   2. Meeting the diagnosis criteria for diabetes
2. History (past 3 years) of hyperparathyroidism, nephrolithiasis or hypercalcemia.
3. Pregnancy (past 1 year by report or positive pregnancy test at screening), intent to become pregnant in the next 4 years or unprotected intercourse. History of gestational diabetes is not an exclusion criterion.
4. Currently breastfeeding.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2423 (Actual)
Dates: Start 2013-10; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anastassios Pittas, MD, MS, Principal Investigator — Tufts Medical Center
Locations (25):
- United States (25):
  - Southwest American Indian Center, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado, Denver, Aurora, Colorado
  - Orlando VA Medical Center, Orlando, Florida
  - Florida Hospital Translational Research Institute, Orlando, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Tulane University Health Sciences, New Orleans, Louisiana
  - Maine Medical Center, Scarborough, Maine
  - MedStar Community Clinical Research Center, Hyattsville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Health Partners Riverside Clinic, Minneapolis, Minnesota
  - Omaha VA Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Beth Israel Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Corbin KD, Pittas AG, Desouza C, Grdinovac KK, Herzig KH, Kashyap SR, Kim SH, Nelson J, Rasouli N, Vickery EM, Knowler WC, Pratley RE. Indices of hepatic steatosis and fibrosis in prediabetes and association with diabetes development in the vitamin D and type 2 diabetes study. J Diabetes Complications. 2023 Jun;37(6):108475. doi: 10.1016/j.jdiacomp.2023.108475. Epub 2023 Apr 12. PMID 37104979
- [Derived] Chatterjee R, Davenport CA, Vickery EM, Johnson KC, Kashyap SR, LeBlanc ES, Nelson J, Dagogo-Jack S, Pittas AG, Hughes BD; D2d Research Group. Effect of intratrial mean 25(OH)D concentration on diabetes risk, by race and weight: an ancillary analysis in the D2d study. Am J Clin Nutr. 2023 Jul;118(1):59-67. doi: 10.1016/j.ajcnut.2023.03.021. Epub 2023 Mar 29. PMID 37001590
- [Derived] Desouza C, Chatterjee R, Vickery EM, Nelson J, Johnson KC, Kashyap SR, Lewis MR, Margolis K, Pratley R, Rasouli N, Sheehan PR, Pittas AG; D2d Research Group. Electronic address: d2d@tuftsmedicalcenter.org. The effect of vitamin D supplementation on cardiovascular risk in patients with prediabetes: A secondary analysis of the D2d study. J Diabetes Complications. 2022 Aug;36(8):108230. doi: 10.1016/j.jdiacomp.2022.108230. Epub 2022 Jun 12. PMID 35753926
- [Derived] Johnson KC, Pittas AG, Margolis KL, Peters AL, Phillips LS, Vickery EM, Nelson J, Sheehan PR, Reboussin D, Malozowski S, Chatterjee R; D2d research group. Safety and tolerability of high-dose daily vitamin D3 supplementation in the vitamin D and type 2 diabetes (D2d) study-a randomized trial in persons with prediabetes. Eur J Clin Nutr. 2022 Aug;76(8):1117-1124. doi: 10.1038/s41430-022-01068-8. Epub 2022 Feb 9. PMID 35140313
- [Derived] Chatterjee R, Fuss P, Vickery EM, LeBlanc ES, Sheehan PR, Lewis MR, Dolor RJ, Johnson KC, Kashyap SR, Nelson J, Pittas AG; D2d Research Group. Vitamin D Supplementation for Prevention of Cancer: The D2d Cancer Outcomes (D2dCA) Ancillary Study. J Clin Endocrinol Metab. 2021 Aug 18;106(9):2767-2778. doi: 10.1210/clinem/dgab153. PMID 33693713
- [Derived] Hsia DS, Rasouli N, Pittas AG, Lary CW, Peters A, Lewis MR, Kashyap SR, Johnson KC, LeBlanc ES, Phillips LS, Hempe JM, Desouza CV; D2d Research Group. Implications of the Hemoglobin Glycation Index on the Diagnosis of Prediabetes and Diabetes. J Clin Endocrinol Metab. 2020 Mar 1;105(3):e130-8. doi: 10.1210/clinem/dgaa029. PMID 31965161
- [Derived] Pittas AG, Dawson-Hughes B, Sheehan P, Ware JH, Knowler WC, Aroda VR, Brodsky I, Ceglia L, Chadha C, Chatterjee R, Desouza C, Dolor R, Foreyt J, Fuss P, Ghazi A, Hsia DS, Johnson KC, Kashyap SR, Kim S, LeBlanc ES, Lewis MR, Liao E, Neff LM, Nelson J, O'Neil P, Park J, Peters A, Phillips LS, Pratley R, Raskin P, Rasouli N, Robbins D, Rosen C, Vickery EM, Staten M; D2d Research Group. Vitamin D Supplementation and Prevention of Type 2 Diabetes. N Engl J Med. 2019 Aug 8;381(6):520-530. doi: 10.1056/NEJMoa1900906. Epub 2019 Jun 7. PMID 31173679
- [Derived] Aroda VR, Sheehan PR, Vickery EM, Staten MA, LeBlanc ES, Phillips LS, Brodsky IG, Chadha C, Chatterjee R, Ouellette MG, Desouza C, Pittas AG; D2d Research Group. Establishing an electronic health record-supported approach for outreach to and recruitment of persons at high risk of type 2 diabetes in clinical trials: The vitamin D and type 2 diabetes (D2d) study experience. Clin Trials. 2019 Jun;16(3):306-315. doi: 10.1177/1740774519839062. Epub 2019 Apr 22. PMID 31007049
- [Derived] LeBlanc ES, Pratley RE, Dawson-Hughes B, Staten MA, Sheehan PR, Lewis MR, Peters A, Kim SH, Chatterjee R, Aroda VR, Chadha C, Neff LM, Brodsky IG, Rosen C, Desouza CV, Foreyt JP, Hsia DS, Johnson KC, Raskin P, Kashyap SR, O'Neil P, Phillips LS, Rasouli N, Liao EP, Robbins DC, Pittas AG; D2d Research Group. Baseline Characteristics of the Vitamin D and Type 2 Diabetes (D2d) Study: A Contemporary Prediabetes Cohort That Will Inform Diabetes Prevention Efforts. Diabetes Care. 2018 Aug;41(8):1590-1599. doi: 10.2337/dc18-0240. Epub 2018 Jun 25. PMID 29941495
- [Derived] Lewis MR, Macauley RC, Sheehan PR, Staten MA, Phillips LS, Rasouli N, Pittas AG; D2d Research Group. Management of Hemoglobin Variants Detected Incidentally in HbA1c Testing: A Common Problem Currently Lacking a Standard Approach. Diabetes Care. 2017 Feb;40(2):e8-e9. doi: 10.2337/dc16-1667. Epub 2016 Nov 29. No abstract available. PMID 27899488
- [Derived] Pittas AG, Dawson-Hughes B, Sheehan PR, Rosen CJ, Ware JH, Knowler WC, Staten MA; D2d Research Group. Rationale and design of the Vitamin D and Type 2 Diabetes (D2d) study: a diabetes prevention trial. Diabetes Care. 2014 Dec;37(12):3227-34. doi: 10.2337/dc14-1005. Epub 2014 Sep 9. PMID 25205139

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Vitamin D (Cholecalciferol)
Started | 1212 | 1211
Completed | 1211 | 1211
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D (Cholecalciferol) | Total
Number analyzed (Participants) | 1212 | 1211 | 2423
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.0) | 59.6 (9.9) | 60.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 545 | 541 | 1086
  Male | 667 | 670 | 1337
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 105 | 120 | 225
  Not Hispanic or Latino | 1107 | 1091 | 2198
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 5 | 13
  Asian | 64 | 66 | 130
  Native Hawaiian or Other Pacific Islander | 0 | 5 | 5
  Black or African American | 315 | 301 | 616
  White | 806 | 810 | 1616
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 24 | 43
Region of Enrollment [Number; unit: participants]
  United States | 1212 | 1211 | 2423
Fasting plasma glucose (mg/dl) [Mean (Standard Deviation); unit: mg/dl] | 107.8 (7.4) | 108.0 (7.4) | 107.9 (7.4)
2-Hr post-load plasma glucose (mg/dl) [Mean (Standard Deviation); unit: mg/dl] | 137.6 (34.3) | 136.9 (34.3) | 137.2 (34.3)
Glycated hemoglobin (%) [Median (Standard Deviation); unit: %] | 5.9 (0.2) | 5.9 (0.2) | 5.9 (0.2)
Serum 25-hydroxyvitamin D (ng/ml) [Mean (Standard Deviation); unit: ng/ml] | 28.2 (10.1) | 27.7 (10.2) | 28.0 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Time to Development of Diabetes
Description: New-onset diabetes was based on annual glycemic testing of fasting plasma glucose, glycated hemoglobin, and 2-hour post-load plasma glucose and semiannual testing of fasting plasma glucose and glycated hemoglobin. If two or three of the glycemic measures met the 2010 ADA thresholds for diabetes, the participant was considered to have met the diabetes outcome. When only the measure for fasting plasma glucose or glycated hemoglobin met the threshold, confirmatory testing was performed for the positive measure within 8 weeks. If only the measure for 2-hour post-load plasma glucose met the threshold, then a 75-g oral glucose tolerance test to reassess all three glycemic measures was repeated. If the repeat measure was positive or both fasting plasma glucose and glycated hemoglobin were positive (in the case of a repeat oral glucose tolerance test), than the participant was considered to have met the diabetes outcome.
Time Frame: Approximately 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D (Cholecalciferol)
Number analyzed (Participants) | 1212 | 1211
Participants | 323 | 293

2. Secondary Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: 25OHD Concentration
Time Frame: Approximately 48 months
Reporting Status: Not Posted

3. Secondary Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: Race (as a Proxy for Skin Pigmentation)
Description: Race and ethnic group were reporting by the participant. The category "other" includes American Indian or Alaska Native; Native Hawaiian or other Pacific Islander; and other race. Ethnic group includes any race.
Time Frame: Approximately 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D (Cholecalciferol)
Number analyzed (Participants) | 1212 | 1211
Participants
  Race: White | 806 | 810
  Race: Black | 315 | 301
  Race: Other | 91 | 100
  Ethnic Group: Hispanic | 105 | 120
  Ethnic Group: Non-Hispanic | 1107 | 1091

4. Secondary Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: Pre-diabetes Criteria (Two vs. Three Criteria)
Description: Participants met at least two of three glycemic criteria for prediabetes: fasting plasma glucose level, 100 to 125 mg per deciliter (5.6 to 6.9 mmol per liter); plasma glucose level 2 hours after a 75-g oral glucose load, 140 to 199 mg per deciliter (7.8 to 11.0 mmol per liter) (impaired glucose tolerance); and glycated hemoglobin level, 5.7 to 6.4% (39 to 47 mmol per mole).
Time Frame: Approximately 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D (Cholecalciferol)
Number analyzed (Participants) | 1212 | 1211
Participants
  Met all three criteria | 429 | 427
  Met two criteria | 783 | 784

5. Secondary Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: BMI
Time Frame: Approximately 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D (Cholecalciferol)
Number analyzed (Participants) | 1212 | 1211
Participants
  <30 | 429 | 435
  ≥30 | 783 | 776

6. Secondary Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: Waist Circumference
Time Frame: Approximately 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D (Cholecalciferol)
Number analyzed (Participants) | 1212 | 1211
Participants
  <Median of 104.2 cm | 585 | 620
  ≥Median of 104.2 cm | 627 | 591

7. Secondary Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: Age
Time Frame: Approximately 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D (Cholecalciferol)
Number analyzed (Participants) | 1212 | 1211
Participants
  25-44 | 103 | 106
  45-59 | 439 | 468
  ≥ 60 | 670 | 637

8. Secondary Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: Geographic Location (as a Proxy for Sun Exposure)
Time Frame: Approximately 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D (Cholecalciferol)
Number analyzed (Participants) | 1212 | 1211
Participants
  At or above 37° north latitude | 898 | 892
  Below 37° north latitude | 314 | 319

9. Secondary Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: Calcium Intake From Supplements
Time Frame: Approximately 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D (Cholecalciferol)
Number analyzed (Participants) | 1212 | 1211
Participants
  No intake | 793 | 826
  Any intake | 419 | 385

10. Secondary Outcome: Blood Plasma 25OHD Concentration.
Time Frame: Approximately 48 months
Reporting Status: Not Posted

11. Secondary Outcome: Number of Participants With Adverse Events.
Time Frame: Approximately 48 months
Reporting Status: Not Posted

12. Secondary Outcome: Change in Blood Pressure as a Continuous Variable.
Time Frame: Approximately 48 months
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants Who Discontinue Study Pills.
Time Frame: Approximately 48 months
Reporting Status: Not Posted

14. Secondary Outcome: Change in FPG as a Continuous Variable.
Time Frame: Every 12 months for approximately 48 months
Reporting Status: Not Posted

15. Secondary Outcome: Change in 2hPG as a Continuous Variable.
Time Frame: Every 12 months for approximately 48 months.
Reporting Status: Not Posted

16. Secondary Outcome: Change in HbA1c as a Continuous Variable.
Time Frame: Every 6 months for approximately 48 months
Reporting Status: Not Posted

17. Secondary Outcome: Measurement of Insulin Resistance (Derived From the OGTT).
Time Frame: Every 12 months for approximately 48 months
Reporting Status: Not Posted

18. Secondary Outcome: Measurement of Beta Cell Secretion (Derived From the OGTT)
Time Frame: Every 12 months for approximately 48 months
Reporting Status: Not Posted

19. Secondary Outcome: Identification of Characteristics Associated With the Variability in Achieved 25OHD Concentration.
Time Frame: Every 12 months for approximately 48 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: Sex
Time Frame: Approximately 48 months.
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: Ethnicity
Time Frame: Approximately 48 months.
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Variability of Response to Vitamin D Supplementation by Baseline Characteristic: 2 Hour Plasma Glucose
Time Frame: Approximately 48 months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Time to Development of Cancer.
Time Frame: Approximately 48 months.
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Time to Development of Cardiovascular Event.
Time Frame: Approximately 48 months.
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Incidence of Cancer in a Pre-diabetes Population Defined by the Modern American Diabetes Association Criteria.
Time Frame: Approximately 48 months.
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Incidence of Cardiovascular Disease in a Pre-diabetes Population Defined by the Modern American Diabetes Association Criteria.
Time Frame: Approximately 48 months.
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Quality of Life and Mood Scores in Pre-diabetes Population Using a Validated Instrument (PROMIS-29 Profile v2.0 and a General Question on Perception of Overall Health From the PROMIS Scale 1.2).
Time Frame: One time assessment at the month 24 visit.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Placebo | Vitamin D (Cholecalciferol)
All-Cause Mortality (participants affected / at risk) | 5/1212 | 5/1211
Serious Adverse Events (participants affected / at risk) | 153/1212 | 173/1211
Other Adverse Events (participants affected / at risk) | 26/1212 | 31/1211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1212) | Vitamin D (Cholecalciferol) (N=1211)
Death (Cardiac disorders) | 5 | 5
Hospitalization (Cardiac disorders) | 148 | 168
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1212) | Vitamin D (Cholecalciferol) (N=1211)
Hypercalcemia (Endocrine disorders) | 3 (3) | 5 (5)
Fasting urine calcium: creatinine ratio >0.375 (Endocrine disorders) | 1 (1) | 1 (1)
Low estimated glomerular filtration rate (Endocrine disorders) | 2 (2) | 1 (1)
Nephrolithiasis (Endocrine disorders) | 20 (21) | 24 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT01942694/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT01942694/SAP_001.pdf